CLINICAL TRIAL: NCT05457660
Title: Transverse Study About QOL for Colostomized or Ileostomized Patients During Their Home Hospitalization
Acronym: STOM'HAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondation Sante Service (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A00014-39
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Colostomy; Ileostomy; Home Hospitalization
Keywords: Home Hospitalization; Colostomy; Ileostomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goalf of the study is to have a basis about QOL for colo-stoma and ileo-stoma for patients which are hospitalized at home. The QOL measurement is done with a questionnaire of several items made by stomatherapist and also using EQ5D QOL form.

After reviewing of the data, our goal is to create or improve some solutions to improve their QOL during their home hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Colo-stomy or Ileo-stomy patient
* Patient hospitalized at home by Fondation Sante Service (Fr)
* 18 YO or more
* Non-opposition to the study

Exclusion Criteria:

* Patient not able to read or properly understand the Information Consent Form and not able to complete the questionnaire for any reason.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stoma : Colostomy and Ileostomy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Measuring the quality of life of colostomized or ileostomized patients in home hospitalization | 4 months

SECONDARY OUTCOMES:
Identify patient issues and needs. | 4 months
Analyze the results by subgroups of patients: according to the type of stoma (ileostomy vs. colostomy; temporary stomy vs. permanent stoma), age of the stoma, age, pathology. | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Santé Service, Levallois-Perret, France

IPD SHARING:
Plan to Share IPD: No